CLINICAL TRIAL: NCT06044623
Title: Implementing Geriatric Assessment for Dose Optimization of CDK 4/6-inhibitors in Older Breast Cancer Patients - a Pragmatic Randomized-controlled Trial (IMPORTANT Trial)
Brief Title: Implementing Geriatric Assessment for Dose Optimization of Cyclin-dependent Kinase (CDK) 4/6-inhibitors in Older Breast Cancer Patients
Acronym: IMPORTANT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Region Örebro County (Other)
Collaborators: University of Patras (Other); University of Florence (Other); Azienda USL Toscana Centro (Other); Helsinki University Central Hospital (Other); Institute for Medical Technology Assessment - the Netherlands (Unknown); Security Labs Consulting Limited (Unknown); Circular Economy Foundation (Unknown); Universidad Nacional de Educación a Distancia (Other); Hellenic Cooperative Oncology Group (Other); University Hospital, Akershus (Other); Uppsala County Council, Sweden (Other Government); Hospital Clinic of Barcelona (Other); Phaze Clinical Research & Pharma Consulting (Unknown); Bröstcancerförbundet (Unknown); Eunomia Ltd (Unknown); University of Applied Sciences and Arts Northwestern Switzerland (Other); CareAcross (Industry); Örebro University, Sweden (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 280232
Record Dates: First submitted 2023-09-13; First posted 2023-09-21 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Breast Cancer; Advanced Breast Cancer; Quality of Life; Toxicity; Older Patients
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Lower initial dose of CDK 4/6-inhibitor (vulnerable/frail patient cohort) (Experimental): -1 level dose reduction as initial dose of either one of the CDK 4/6-inhibitors: Palbociclib 100 mg x 1 for 21 days with 7 days off; or Ribociclib 400 mg x 1 for 21 days with 7 days off; or Abemaciclib 100 mg x 2 daily added to endocrine therapy.
  Interventions: Drug: CDK 4/6 inhibitors; Drug: Endocrine therapy
- Full initial dose of CDK 4/6-inhibitor (vulnerable/frail patient cohort) (Active Comparator): Full initial dose of either one of the CDK 4/6-inhibitors: Palbociclib 125 mg x 1 for 21 days with 7 days off; or Ribociclib 600 mg x 1 for 21 days with 7 days off; or Abemaciclib 150 mg x 2 daily) added to physician's choice endocrine therapy.
  Interventions: Drug: CDK 4/6 inhibitors; Drug: Endocrine therapy
- Full initial dose of CDK 4/6-inhibitor (fit patient cohort) (Other): Full initial dose of either one of the CDK 4/6-inhibitors: Palbociclib 125 mg x 1 for 21 days with 7 days off; or Ribociclib 600 mg x 1 for 21 days with 7 days off; or Abemaciclib 150 mg x 2 daily) added to physician's choice endocrine therapy.
  Interventions: Drug: CDK 4/6 inhibitors; Drug: Endocrine therapy

INTERVENTIONS:
Drug: CDK 4/6 inhibitors — Either Palbociclib, Ribociclib or Abemaciclib
Drug: Endocrine therapy — Either Letrozole, Anastrozole, Exemestane or Fulvestrant in combination with CDK 4/6-inhibitor

SUMMARY:
IMPORTANT study is a multicenter, open-label, prospective, randomized-controlled, non-inferiority trial with a pragmatic approach involving older patients (≥ 70 years old) with advanced hormone receptor (HR)-positive/human epidermal growth factor receptor 2 (HER2)-negative breast cancer, not amenable for curative treatment and without prior therapy for advanced disease, who are suitable to receive CDK 4/6-inhibitors plus endocrine therapy as first line therapy. The study implements two approaches with high level of evidence, namely the use of comprehensive geriatric assessment (CGA) approach in treatment decision making and the use of CDK 4/6-inhibitors as the initial treatment of choice, to investigate whether a common clinical practice (starting dose reduction of CDK 4/6-inhibitors in older patients) with evidence of low certainty can be standardized using a more individualized-based approach.

On the basis of baseline CGA assessment, patients will either receive full dose of CDK 4/6-inhibitors plus endocrine therapy (if patients are fit according to CGA) or be randomized to full dose vs. reduced initial dose of CDK 4/6-inhibitors (if vulnerable or frail according to CGA). The study hypothesis is that adjusting the dose according to vulnerability will allow patients to tolerate treatment better without jeopardizing the treatment efficacy.

This project has received funding from the European Union's HORIZON 2022 research and innovation actions supporting the implementation of the Mission on Cancer under grant agreement No 101104589.

ELIGIBILITY:
Inclusion Criteria:

The following inclusion criteria will be applied:

1. Patients male or female aged at least 70 years old at the time of informed consent.
2. Histologically or cytologically confirmed diagnosis of HR-positive (defined as estrogen-receptor ≥ 1%), HER2-negative breast cancer according to analysis of the most recent tumor specimen by local laboratory.
3. Advanced (locoregionally recurrent or metastatic) breast cancer not amenable to curative treatment.
4. No prior systemic treatment for advanced disease (recurrence during neo-/adjuvant endocrine therapy is allowed). A prior period of treatment with aromatase inhibitors or fulvestrant for up to 28 days from the CDK 4/6-inhibitor initiation is allowed.
5. Adjuvant treatment with CDK 4/6-inhibitors is allowed provided a disease-free interval from treatment end >12 months.
6. Either measurable disease or non-measurable bone only disease, but evaluable according to RECIST criteria 1.1.
7. Written informed consent prior to any study-specific procedures.
8. Adequate organ function as defined in the summary of product characteristics (SmPC) for the CDK 4/6-inhibitors that is planned to be used.
9. Able to swallow capsules.
10. Able to understand and consent in English language or in native language for each participating country.

Exclusion Criteria:

Eligible patients will be excluded if they have one of the following criteria:

1. Patients considered from treating physician as non-suitable for treatment with CDK 4/6-inhibitors.
2. Contraindications according to SmPC for the CDK 4/6-inhibitors that is planned to be used.
3. Presence of visceral crisis, lymphangitis carcinomatosis, or leptomeningeal carcinomatosis.
4. History of any other cancer (except of non-melanoma skin cancer or carcinoma in-situ of the cervix), unless in complete remission with no therapy for a minimum of 3 years.
5. Participating in other interventional trial.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 495 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2028-10-31 (Estimated); Study Completion 2029-05-31 (Estimated)

PRIMARY OUTCOMES:
Time to treatment failure | Up to 5 years from treatment initiation
  The time from randomization to treatment discontinuation because of any reason including disease progression, treatment toxicity, or death due to any cause.

SECONDARY OUTCOMES:
Overall treatment utility (OTU) | Three months after treatment initiation
  A composite endpoint that will be assessed at the first efficacy evaluation. OTU incorporates objective and participant-reported outcome measures of anticancer efficacy, tolerability and acceptability of treatment providing a simple "good, intermediate or poor" categorization of outcome.
Overall survival | Up to 5 years from treatment initiation
  The time from randomization to death from any cause.
Progression free survival | Up to 5 years from treatment initiation
  The time from randomization to first documented evidence of disease progression or death from any cause.
Time to chemotherapy initiation | Up to 5 years from treatment initiation
  The time from randomization until the initiation of chemotherapy at any treatment line after CDK 4/6-inhibitors.
Frequency of adverse events | Up to 5 years from treatment initiation
  Adverse events will be assessed based on adverse events, as graded by CTCAE v 5.0 before each cycle and up to 28 days after the end of CDK 4/6-inhibitors.
Assessment of Quality of life | Until disease progression, participant / physician decision to stop, death, or up to 24 months from treatment initiation whichever occurs first
  Quality of life will be assessed using three validated questionnaires, EORTC Quality of Life Questionnaire (QLQ)-C30, Elderly (ELD)-14, and European Quality of Life-5 Dimensions-5 Levels (EQ-5D-5L).
Time until Quality of life deterioration | Until disease progression, participant / physician decision to stop, death, or up to 24 months from treatment initiation whichever occurs first
  QoL deterioration, defined as the time from randomization until any clinically meaningful worsening (using minimal important differences as cut-off) of any QoL aspect measured by the questionnaires.
Cost effectiveness | Up to 24 months from treatment initiation
  Resource use, length of life and quality of life data will be collected during the trial for the purpose of conducting an economic evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Antonios Valachis, Assoc Prof, Study Chair — Region Örebro län
Locations (12):
- Department of Oncology, Helsinki University Hospital Comprehensive Cancer Center and University of Helsinki, Helsinki, Finland
- Greece (5):
  - Fourth Oncology Department & Comprehensive Clinical Trials Center, Metropolitan Hospital, Athens
  - Second Department of Medical Oncology, Hygeia Hospital, Athens
  - Division of Oncology, Department of Medicine, University Hospital, University of Patras Medical School, Pátrai
  - Medical Oncology Unit, S. Andrew Hospital, Pátrai
  - Second Department of Medical Oncology, Euromedica General Clinic, Thessaloniki
- Italy (2):
  - Radiation Oncology Unit - Oncology Department, Azienda Ospedaliero Universitaria Careggi, Florence
  - "Sandro Pitigliani" Department of Medical Oncology, Hospital of Prato, Prato
- Department of Oncology, Akershus University Hospital (AHUS), Oslo, Norway
- Department of Medical Oncology, Hospital Clinic of Barcelona, Barcelona, Spain
- Sweden (2):
  - Department of Oncology, Örebro University Hospital, Örebro
  - Department of Oncology, Uppsala University Hospital, Uppsala

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Valachis A, Biganzoli L, Christopoulou A, Fjermeros K, Fountzila E, Geisler J, Gomez-Bravo R, Karihtala P, Kosmidis P, Koutras A, Linardou H, Lindman H, Martinez-Ballestero I, Rodriguez AB, Meattini I, Munoz-Mateu M, Othman M, Psyrri A, Risi E, Schiza A, Spathas N, Utriainen M, Visani L, Ballesteros S, Basdekis I, Hay SD, Fotis T, Fricker S, de Graaf G, Jenset M, Kanters T, Lampropoulos K, Markou C, Mastoraki K, Nanou C, Reales Aviles JM, Santaholma M, Kosmidis T. Implementing geriatric assessment for dose optimization of CDK4/6 inhibitors in older breast cancer patients. Future Oncol. 2024;20(37):2937-2948. doi: 10.1080/14796694.2024.2413841. Epub 2024 Oct 21. PMID 39431459